CLINICAL TRIAL: NCT05941923
Title: A Respiratory Critical Care Nurse Training Program for Countries Without Registered Respiratory Therapist: A Randomize Clinical Trial
Brief Title: Respiratory Critical Care Nurse Training Program
Acronym: RCCN Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Principal Investigator, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Respiratory Nurse
Record Dates: First submitted 2023-06-22; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Morality; Treatment Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical superiority trial with two-arm parallel group design
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple blinding : Patients, respiratory critical care nurses, and data analyzers will be blinded to the allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group, who will receive specialized respiratory care from RCCN from the time they arrive in the emergency room until their discharge from the hospital
  Interventions: Other: respiratory critical care support
- Control group (No Intervention): No intervention group, who will receive only routine care without any intervention.

INTERVENTIONS:
Other: respiratory critical care support — Patients in the intervention group will be received respiratory critical care support
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial study is to evaluate the clinical effectiveness of respiratory critical care nurses (RCCN) in improving outcomes for critically ill patients who require admission to the intensive care units (ICUs). The main question it aims to answer is: What is the effect of the respiratory critical care nurse in improving outcomes for critically ill patients? Participants will consist of critically ill patients who will be randomly allocated in a 1:1 ratio into two groups: the intervention group, who will receive specialized respiratory care from RCCN from the time they arrive in the emergency room until their discharge from the hospital, and the control group, who will receive only routine care.

DETAILED DESCRIPTION:
A randomized controlled clinical superiority trial with triple blinding and a two-arm parallel group design will be conducted at Baqiyatallah University of Medical Sciences in Tehran, Iran between November 22, 2023, and November 10, 2024. The aim of this study will to evaluate the clinical effectiveness of respiratory critical care nurses (RCCN) in improving outcomes for critically ill patients who require admission to the intensive care units (ICUs). Participants will consist of critically ill patients who will be randomly allocated in a 1:1 ratio into two groups: the intervention group, who will receive specialized respiratory care from RCCN from the time they arrive in the emergency room until their discharge from the hospital, and the control group, who will receive only routine care

ELIGIBILITY:
Inclusion Criteria:

* They are at least 18 years old,
* Critically ill patients who need critical care,
* They have no history of heart disease, stroke, autoimmune disease, neuromuscular diseases, cancer, or cardio-respiratory arrest,
* They are willing to participate in the study.

Exclusion Criteria:

* Patients with pregnancy and breastfeeding women
* Patients at end-stage medical condition
* Patients with planned withdrawal of treatment

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | through study completion, an average of 3 months
  The primary outcome of this study will be to compare mortality rates between two study groups.

SECONDARY OUTCOMES:
Treatment failures | through study completion, an average of 3 months
  The secondary outcome will be the proportion of treatment failures, which is defined by a composite endpoint consisting of the need for non-invasive ventilation (NIV), intubation, or death

OTHER OUTCOMES:
Rate of endotracheal intubation | through study completion, an average of 3 months
  Rate of endotracheal intubation will be compare between two study groups
Rate of non-invasive ventilation (NIV) | through study completion, an average of 3 months
  Rate of non-invasive ventilation (NIV) will be compare between two study groups
Rate of ventilator-associated pneumonia (VAP) | through study completion, an average of 3 months
  Rate of ventilator-associated pneumonia (VAP) will be compare between two study groups
Rate of a two-point decrease based on the clinical World Health Organization (WHO) scale | through study completion, an average of 3 months
  These changes will be measured from randomization to ICU discharge, which is defined as continuous and uneventful improvement without requiring additional respiratory support, from the date of inclusion until a two-point decrease in the clinical WHO scale. The clinical WHO measures the severity of a patient's hospitalization status on a seven-point ordinal scale as follows: (a) not hospitalized, capable of resuming normal activities, (b) not hospitalized but unable to resume normal activities, (c) hospitalized, no oxygen therapy, (d) hospitalized and requiring oxygen therapy, (e) hospitalized and requiring NIV or nasal high-flow oxygen, (f) hospitalized and requiring mechanical ventilation, (g) hospitalized and requiring mechanical ventilation (MV) with other organ support (vasopressors, renal replacement therapy, extracorporeal life support), and (h) dead.
Pre-ICU length of stay | through study completion, an average of 3 months
  Pre-ICU length of stay in days will be compare between two study groups
ICU length of stay | through study completion, an average of 3 months
  ICU length of stay in days will be compare between two study groups
Post-ICU length of stay | through study completion, an average of 3 months
  Post-ICU length of stay in days will be compare between two study groups
Functional oxygen saturation (SaO2) | through study completion, an average of 3 months
  SaO2 will be measured through an arterial blood gas (ABG) analysis and compare between two study groups
partial pressure of oxygen (PaO2) | through study completion, an average of 3 months
  PaO2 will be measured through an arterial blood gas (ABG) analysis and compare between two study groups
Oxygen saturation SpO2 | through study completion, an average of 3 months
  SpO2 will be measured noninvasive using a pulse oximeter and compare between two study groups